CLINICAL TRIAL: NCT00126074
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel Design Study to Evaluate the Efficacy and Safety of Intravenous Tedisamil Sesquifumarate in the Rapid Conversion to Normal Sinus Rhythm in Female Subjects With Recent Onset Atrial Fibrillation or Flutter
Brief Title: Intravenous Tedisamil in the Rapid Conversion of Atrial Fibrillation or Flutter to Normal Sinus Rhythm in Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S219.3.118; 2004-000346-21
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2006-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial fibrillation, atrial flutter, anti-arrhythmic agents, conversion to normal sinus rhythm
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

INTERVENTIONS:
Drug: Tedisamil sesquifumarate

SUMMARY:
The purpose of this study is to demonstrate the ability of tedisamil to convert atrial fibrillation or flutter into normal sinus rhythm (NSR) in female patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign informed consent before screening examinations are performed and before the study drug is administered
* Females > 18 years of age
* Subjects with documented (60 second rhythm strip) symptomatic atrial fibrillation or flutter (duration > 3 hours and < 45 days) at the time of randomization
* Subjects who are in no distress and hemodynamically stable (supine systolic blood pressure > 90 mmHg and diastolic blood pressure < 105 mmHg)

Exclusion Criteria:

* Pregnancy and lactation
* Acute myocardial infarction and cerebrovascular accidents
* Coronary syndromes and congestive heart failure (CHF) New York Heart Association (NYHA) IV
* Life-threatening ventricular arrhythmias and electrocardiogram (ECG) abnormalities
* Concurrent antiarrhythmic treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (26):
- United States (2):
  - Site 26, Honolulu, Hawaii
  - Site 27, Tullahoma, Tennessee
- Bulgaria (6):
  - Site 5, Pleven
  - Site 2, Sofia
  - Site 3, Sofia
  - Site 4, Sofia
  - Site 6, Sofia
  - Site 7, Sofia
- Site 8, Mannheim, Germany
- Hungary (7):
  - Site 11, Budapest
  - Site 12, Budapest
  - Site 14, Budapest
  - Site 15, Budapest
  - Site 9, Budapest
  - Site 13, Kecskemét
  - Site 10, Korhaz
- Site 16, Piacenza, Italy
- Poland (9):
  - Site 22, Chrzanów
  - Site 20, Gdansk
  - Site 25, Gdynia
  - Site 19, Katowice
  - Site 18, Krakow
  - Site 24, Szczecin
  - Site 17, Tarnów
  - Site 23, Wałbrzych
  - Site 21, Zakopane